CLINICAL TRIAL: NCT05705596
Title: Einfluss Des süßmodulierenden Polyphenols Hesperetin in Kombination Mit Saccharose Auf Die Blutglukose-Regulierung Und Energieaufnahme in Abhängigkeit Der Süßwahrnehmung
Brief Title: Impact of Hesperetin in Combination With Sucrose on Energy Metabolism
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Barbara Lieder, Professor and Vice Chair Department of Physiological Chemistry, University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 706014-2
Record Dates: First submitted 2023-01-17; First posted 2023-01-31 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Blood Glucose Fluctuations; Hunger
MeSH Terms: interventions — Sucrose; Dietary Sucrose; hesperetin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sucrose (Experimental): 10% (w/v) sucrose in water
  Interventions: Other: Sucrose
- Hesperetin (Experimental): 7% (w/v) sucrose in water + 50 mg/L Hesperetin
  Interventions: Drug: Hesperetin

INTERVENTIONS:
Other: Sucrose — 10% sucrose corresponding to a regular soft drink
  Other Names: table sugar
  Arms: Sucrose
Drug: Hesperetin — increases sweetness of 7% sucrose solution to match sweetness of 10% sucrose solution
  Other Names: (2S)-3',5,7-Trihydroxy-4'-methoxyflavan-4-one; CAS number 520-33-2
  Arms: Hesperetin

SUMMARY:
The aim of this cross-over intervention study is to investigate the influence of the sweet-modulating substance hesperetin in combination with sucrose in comparison to an equally sweet-tasting sucrose-only solution on markers of energy metabolism.

DETAILED DESCRIPTION:
The study is designed as a randomised cross-over intervention study with two arms. The aim is to investigate the influence of a 10% sucrose solution, corresponding to the sugar content of a conventional soft drink, compared to an equally sweet-tasting 7% sucrose solution in combination with 50 mg/L of the polyphenol hesperetin, on time-dependent blood glucose fluctuations and ad libitum energy intake in metabolically healthy male volunteers.

To investigate the underlying mechanisms, the individual appetite score, metabolic and hormonal responses to the interventions and circulating extracellular vesicles and their miRNA composition will be measured. In addition, the participants' individual thresholds for sweet taste, preference and consumption for sweet-tasting foods such as sugar and sweeteners, and their body composition will be recorded as potential influencing factors.

ELIGIBILITY:
Inclusion Criteria:

* male
* healthy
* non-smoking
* normal taste responses towards sweet taste

Exclusion Criteria:

* female
* regular smokers
* disturbed glucose and/or lipid metabolism
* regular intake of medication
* known allergies against one of the test compounds
* ageusia
* alcohol or drug addiction
* intake of antibiotics within the past 2 months

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose concentration | 15, 30, 60, 90, and 120 minutes after drinking the test solution
  Change compared to baseline in blood glucose concentration [mg/dL] in plasma samples after drinking the test solution
Change in appetite score | Difference between before and 120 minutes after drinking of the test solution
  Change compared to baseline in the subjective rating of the individual feeling of hunger, fullness, as well as appetite for a snack or for something sweet on a digital visual analog scale in comparison to baseline
Change in food intake | 120 minutes after drinking of the test solution
  Ad libitum food intake from a standardized breakfast

SECONDARY OUTCOMES:
Change in blood glucose regulating hormones | 15, 30, 60, 90, and 120 minutes after drinking the test solution
  Change compared to baseline in Insulin, Glucagon-like peptide 1, and Gastric inhibitory polypeptide concentrations [mmol/L] in plasma samples after drinking the test solution
Change in satiety hormones | 15, 30, 60, 90, and 120 minutes after drinking the test solution
  Change compared to baseline in Polypeptide Y, grehlin, cholecystokinin, and serotonin concentrations [mmol/L] in plasma samples after drinking the test
Change in circulating miRNA | 15, 30, 60, 90, and 120 minutes after drinking the test solution
  Change compared to baseline in circulating extracellular vesicles and their miRNA composition

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lieder, PhD, Principal Investigator — University of Vienna
Locations (1):
- Christian Doppler Laboratory for Taste Research, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaider M, Kimmeswenger I, Schmidt J, Thines C, Wu A, Stoffl TK, Rust P, Ley JP, Krammer GE, Somoza V, Lieder B. Sucrose reduction with maintained sweetness level lowers glycemic fluctuations and energy intake in healthy males. Front Nutr. 2025 Nov 3;12:1682297. doi: 10.3389/fnut.2025.1682297. eCollection 2025. PMID 41256921